CLINICAL TRIAL: NCT04387968
Title: Epidemiological Study of the Covid-19 Presto Test Among Agents of the Local Authorities of CCTVL, Region Centre Val de Loire and Orleans Métropole. Correlation of IgM Level According to Contact With the Public
Brief Title: Epidemiological Study of the Covid-19 Presto Test - The "COVIDOR" Study
Acronym: COVIDOR
Status: Completed | Type: Observational
Sponsor: Raphael Serreau (Other)
Collaborators: François Rabelais University (Unknown); Assistance Publique - Hôpitaux de Paris (Other); University Hospital, Paris (Other)
Responsible Party: Sponsor-Investigator, Raphael Serreau, Dr Raphaël SERREAU (PH), Orléans Métropole Service de Médecine Préventive
Organization: Orléans Métropole Service de Médecine Préventive (Other)
Other Study IDs: 2020-A01414-35
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Coronavirus Infection
Keywords: covid-19; serology; depistage; public health; voluntary agents
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood drop to test IgM and IgG by an immunoserology rapid screening autotest and antigenic test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- agents in contact with the public: patients working with children, policemen, desk office
  Interventions: Diagnostic Test: Covid-19 presto test
- agents with no contact with the public: administrative workers
  Interventions: Diagnostic Test: Covid-19 presto test

INTERVENTIONS:
Diagnostic Test: Covid-19 presto test — Use an auto-test in 15 minutes get the results about covid-19 anticorps
  Other Names: Covid-19 viro

SUMMARY:
The "COVIDOR" epidemiological study. Our study would be the first at the community level in Orleans Métropole, aiming to determine the link between a positive IgM level on the serological test and a healthy carrier of covid-19 in agents in contact with the public. It would provide epidemiological surveillance of anti-covid-19 immunity in the community

DETAILED DESCRIPTION:
The metropolitan area of Orléans Métropole has 6,700 agents divided into 250 different trades and consequently multiple exposures and risks.

The global covid-19 pandemic has affected France and the Loiret, the sarscov-2 coronavirus, has infected several thousand people. On May 7, 2020, there were 75 deaths at the CHRO hospital in Orleans, excluding EHPAD. The contamination rate of the population of the Loiret department has been estimated at 5.6% of the population by Public Health France. This rate is very low and does not allow the use of serological screening tests because of too many false positives or false negatives, there should be a prevalence of the disease greater than 60%. The French health authorities do not recommend the use of a screening test at the present time in view of the uncertainties of the results of this test. The Loiret Management Center, the Department and Orléans Métropole have decided to offer a covid-19 serological screening test, the covid-19 presto test, to voluntary territorial agents regardless of their return to work following the national "deconfinement "on May 11, 2020 This can only be done through an epidemiological surveillance study validated as part of a research protocol.

ELIGIBILITY:
Inclusion Criteria:

* All the agents of the 3 local authorities (Loire Valley Region, CCTVL and Orléans Métropole) being voluntary to be tested for the COVID-PRESTO® test COVID-19 IgG / IgM rapid test (whole blood / serum / plasma) - Cassette
* Volunteer to get tested

Exclusion Criteria:

* Opposition to the participation of the study
* Covid-19 disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Blood sample to be taken after self-bite. A consent form is given to the officer.
  A drop of blood is deposited on a coverslip, 2 drops of reagents allow migration to the gel.
  Reading in 15 minutes
  1. strip: negative result
  2. bands: positive result
  An authorized person, subject to medical confidentiality, reports the result in the medical file and informs the agent of the result.
  He is given a paper document signed by the SMP with the procedure to follow.
Sampling Method: Non-Probability Sample
Enrollment: 3228 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Study the prevalence of Covid-19 infection, coronavirus (SARS coronavirus-2) in territorial agents in the 3 structures : CCTVL, Loire Valley Region Centre, Orleans Metropolitan city | 15 minutes
  Covid-19 attack rate by measuring the frequency of anti-covid-19 IgM in each of the territorial structures

SECONDARY OUTCOMES:
Determine if there is a relationship between the profession carried out by the agents of the territorial community of Orleans metropolitan city, the Loire Valley Region, the CCTVL and contamination by covid-19 | 6 months
  Search for a correlation of covid-19 immunity based on the officer's position, if he is in contact with the public.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Raphael SERREAU, MD, PhD, Principal Investigator — Orleans Metropole
Locations (2):
- France (2):
  - Unité de Recherche PARADICT-O - Orléans, Orléans
  - Unité de Recherche PARADICT-O - Service de Médecine - Orléans Métropole, Orléans

IPD SHARING:
Plan to Share IPD: Undecided
Blood sample to be taken after self-bite. A consent form is given to the officer.
  A drop of blood is deposited on a coverslip, 2 drops of reagents allow migration to the gel.
  Reading in 15 minutes
  1. strip: negative result
  2. bands: positive result
  An authorized person, subject to medical confidentiality, reports the result in the medical file and informs the agent of the result.
  He is given a paper document signed by the SMP with the procedure to follow.

REFERENCES:
- [Derived] Hanane G, Amine Z, Roomila N, Prazuck T, Amirouche A, Olivier V, Benyamina A, Serreau R. COVID-19 seroprevalence among local authority workers from Orleans Metropole, the Community of Communes of the Terres du Val de Loire, the local public service management centre of the Loiret department and the Region Centre Val de Loire: a prospective epidemiological study. BMJ Open. 2023 May 22;13(5):e066504. doi: 10.1136/bmjopen-2022-066504. PMID 37217267